CLINICAL TRIAL: NCT06672744
Title: Comparison of the Efficacy of Kinesiotaping and Myofascial Release Techniques in the Treatment of Superior Cluneal Nerve Entrapment Syndrome: A Randomised Single Blind Controlled Trial
Brief Title: Superior Cluneal Nerve Entrapment Syndrome, Kinesiotaping and Myofascial Release Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Savaş Karpuz (Other Government)
Responsible Party: Sponsor-Investigator, Savaş Karpuz, Associate Professor, Konya Beyhekim Training and Research Hospital
Organization: Konya Beyhekim Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Superior Cluneal Nerve Entrapment
MeSH Terms: interventions — Exercise; Muscle Stretching Exercises; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise (Active Comparator): Lumbar muscles (especially quadratus lumborum) and thoracolumbar fascia stretching exercises and strengthening exercises for the lumbar and abdominal muscles were described by the physiotherapist. Participants were asked to perform the exercises three times a day, five days a week.
  Interventions: Other: Exercise
- kinesiotaping (Experimental): Kinesiotaping was performed by the same researcher (XX) for two sessions per week for four weeks with fascia correction technique. The procedure was performed with the participant lying in the prone position. The tape was glued just below the beginning of the iliac crista without stretching. Submaximal tension was continued on the skin in line with the lower fibres of the quadratus lumborum muscle and thorocolumbar fascia. It was terminated without tension at the lower costal fold. I band was applied perpendicular to the line of insertion of the quadratus lumborum and thorocolumbar fascia to the crista iliaca with 50% tension in the middle section without tension at the beginning and end.
  Interventions: Other: Kinesiotaping
- Myofascial release technique (Experimental): Myofascial release technique was applied by the same researcher (YY) twice a week for four weeks. Ischaemic compression was applied to palpable trigger points on the quadratus lumborum muscle. One hand was placed on the inferior crista iliaca and the other hand on the superior inferior costal fold and waited for 3 minutes with minimal tension. The hand was made into a fist and minimal pressure was applied with the proximal phalanges over the quadratus lumborum and the participant was asked to contract and release the muscle for 3 minutes.
  Interventions: Other: Myofascial release technique

INTERVENTIONS:
Other: Exercise — Lumbar muscles (especially quadratus lumborum) and thoracolumbar fascia stretching exercises and strengthening exercises for the lumbar and abdominal muscles were described by the physiotherapist. Participants were asked to perform the exercises three times a day, five days a week
  Other Names: stretching exercises; strengthening exercises
  Arms: exercise
Other: Myofascial release technique — Myofascial release technique was applied by the same researcher (YY) twice a week for four weeks.
  Arms: Myofascial release technique
Other: Kinesiotaping — Kinesiotaping was performed by the same researcher (XX) for two sessions per week for four weeks with fascia correction technique
  Arms: kinesiotaping

SUMMARY:
Myofascial release techniques and/or kinesiotaping may be effective in the treatment of superior cluneal nerve impingement syndrome ?

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with superior cluneal nerve entrapment syndrome

Exclusion Criteria:

* those with communication problems
* those who also described pain in the mid-lumbar region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Visual Analoque Scale | Before treatment, immediately after treatment, 1 month after the end of treatment
  Visual Analoque Scale is a scale consisting of a single 10 cm line and assesses the intensity of pain. Patients were asked to rate the level of pain after being informed that the beginning point on the scale represented no pain and the end point represented the most excruciating pain they had ever experienced
The Roland-Morris Disability Questionnaire | Before treatment, immediately after treatment, 1 month after the end of treatment
  The Roland-Morris Disability Questionnaire is a questionnaire developed to assess functional disabilities in patients with low back pain [15]. In the questionnaire consisting of 24 sentences about functional disabilities, patients are asked to answer each sentence as yes if it fits their situation and no if it does not. Yes answers are calculated as '1' and no answers as '0' points, resulting in a total score between 0-24, with a higher score indicating more disability.

SECONDARY OUTCOMES:
SF-36 Quality of Life Scale | Before treatment, immediately after treatment, 1 month after the end of treatment
  SF-36 Quality of Life Scale is a general quality of life scale frequently used in clinical research. The scale consists of 36 items, which measure 8 different dimensions: physical functions, social functions, role inhibition due to physical problems, physical pain, mental health, role inhibition due to emotional problems, life energy, general health perception. The subscales assess health on a scale of 0 to 100, with higher scores indicating good health quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Training and Research Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Draghici NC, Bolchis R, Popa LL, Vacaras V, Ilut S, Bashimov A, Domnita DM, Dragos HM, Vlad I, Muresanu DF. Rare entrapment neuropathies of the lower extremity: A narrative review. Medicine (Baltimore). 2024 Aug 30;103(35):e39486. doi: 10.1097/MD.0000000000039486. PMID 39213217